CLINICAL TRIAL: NCT05544188
Title: Occurrence and Characteristics of Functional Pathologies of the Musculoskeletal System in Physiotherapy Students and the Possibility of Influencing Them
Brief Title: Functional Pathologies of the Musculoskeletal System in Physiotherapy Students
Acronym: FUNPAMUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kamila Řasová, doc. PhDr. Kamila Řasová, Ph.D., principal investigator, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 29072022
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain, Postural
Keywords: Trigger Point Pain, Myofascial; Motor Activity; Physiotherapy
MeSH Terms: conditions — Low Back Pain; Myofascial Pain Syndromes; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- individual outpatient physiotherapy (Experimental): individual outpatient physiotherapy (7 times in two and a half months, approx. 90 minutes) aimed at correcting functional pathologies of the musculoskeletal system assessed by differential diagnosis (removal of trigger points, stretching of shortened muscles and mobilization of joint blockages) and changing of motor program that led to the occurrence of the functional disorder by means of Motor Programmes Activating Therapy
  Interventions: Diagnostic Test: Differential diagnostic
- Without changing the current habits (Active Comparator): It will not change the existing habits. At the same time, however, these are physiotherapy students who will participate in the classes. Their motor behaviour can thus be influenced in a natural way.
  Interventions: Diagnostic Test: Differential diagnostic

INTERVENTIONS:
Diagnostic Test: Differential diagnostic — Physiotherapy aimed at correcting functional pathologies of the musculoskeletal system assessed by differential diagnosis (removal of trigger points, stretching of shortened muscles and mobilization of joint blockages)

SUMMARY:
This study map the occurrence of functional pathologies of the musculoskeletal system in students of the bachelor's program of physiotherapy of the Third Faculty of Medicine, Charles University, and aim on improvement of them.

DETAILED DESCRIPTION:
The aim of this study is to map the occurrence of functional pathologies of the musculoskeletal system in students of the bachelor's program of physiotherapy of the Third Faculty of Medicine, Charles University, and to examine their postural functions. Another goal is to teach the students of the experimental group how to remove functional pathologies of the musculoskeletal system and how to change their motor behaviour and postural functions so that the development of functional disorders no longer occurs.

ELIGIBILITY:
Inclusion Criteria:

* Bachelor's study of physiotherapy at the Third Faculty of Medicine, Charles University
* The presence of functional pathologies of the musculoskeletal system (verification by means of Trigger Points)

Exclusion Criteria:

* Serious cardiovascular or orthopedic dysfunction
* Neurological disease
* Reduced cognitive functions complicating examination and subsequent therapy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Changes in Trigger Points at 3 months | Pre-assessment (baseline testing), Post-assessment (immediately after the end of three months).
  Local hypertonic change in muscle function arising as a manifestation of pathogenic tension, 0 no trigger point, 2 maximal tiger point (higher value, worse function)

SECONDARY OUTCOMES:
Change in the Foot posture index at 3 and 15 month | Pre-assessment (baseline testing), Post-assessment (immediately after the end of three months), Follow up (at 15 months).
  Clinical examination of the foot type ranging from significantly pronated (values 6 - 12) to significantly supinated (values from -1 to -12) one according to the 6-item, higher value (both negative or positive) means worse function.
Change in Foot morphology and flexibility at 3 and 15 month | Pre-assessment (baseline testing), Post-assessment (immediately after the end of three months), Follow up (at 15 months).
  examination by means of the full foot 3D scanner Footscan® and the software 3D scanner 7.7 while sitting and standing still. Arch high index defines two kinds of pathologies: hypermobility under 0,6, norm 0,7 - 0,8, rigidity 0,9 - 1,3
Change in Postural stability at 3 and 15 month | Pre-assessment (baseline testing), Post-assessment (immediately after the end of three months), Follow up (at 15 months).
  evaluation of the level of postural stability using the total path of displacement of the centre of pressure of the body on the mat in mm and the maximum displacement obtained in the latero-lateral and in the anteroposterior direction in mm (lower number means better function), measurement using the RS Footscan® tensiometric plate, higher value means worse function.
Change in the subtalar joint flexibility at 3 and 15 month | Pre-assessment (baseline testing), Post-assessment (immediately after the end of three months), Follow up (at 15 months).
  mobility of the subtalar joint during the initial phase of walking (software evaluation after walking barefoot on the Footscan® tensiometric plate). Under 5.5° means normal range of pronation and normal function. Higher values mean worse function and pathologic pronation during initial phase of gait.
Change in the foot progression angle at 3 and 15 month | Pre-assessment (baseline testing), Post-assessment (immediately after the end of three months), Follow up (at 15 months).
  rotation of the foot during walking (software evaluation after walking barefoot on the Footscan® tensiometric plate). Normal angle 0-5.4°, in-toeing (inwards rotation) under 0°, out-toeing (outward rotation) above 5.5°.

CONTACTS AND LOCATIONS:
Overall Officials: Kamila Rasova, Principal Investigator — Third Faculty of Medicine
Locations (1):
- Department of rehabilitation, Third Faculty of Medicine, Prague, Czechia